CLINICAL TRIAL: NCT03853967
Title: Lung Cancer Screening by Low Dose CT Scan in a French Department (DEP KP80)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier d'Abbeville (Other)
Responsible Party: Principal Investigator, Olivier LELEU, Head of pneumology department, Centre Hospitalier d'Abbeville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 160048-B81
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Lung Cancer Screening
Keywords: low dose CT scan

STUDY DESIGN:
Intervention Model Description: prospective single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- screening (Experimental): participants performed lung cancer screening by Low Dose CT scan
  Interventions: Other: Low dose CT scan

INTERVENTIONS:
Other: Low dose CT scan — low dose CT scan

SUMMARY:
Lung cancer is the leading cause of cancer death worldwide. The aims of this study were to assess the feasibility and effectiveness of a lung cancer screening pilot program with LD CT scan in a French department (Somme).

DEP KP80 was a single-arm, prospective study started in May 2016. The inclusion criteria were those of the National Lung Screening Trial. An annual LD CT scan was scheduled and 2 rounds were planned. Smoking cessation was encouraged as part of the protocol.

Subjects were selected by General Practitioner or Pneumologist who checked the inclusion criteria and prescribed the CT scan.

DETAILED DESCRIPTION:
Scientific context :

Lung cancer is the deadliest cancer in France and in the world. With around 39500 new cases in 2012 in France, lung cancer ranks fourth regarding cancer incidence for both women and men. In 2012 it caused the highest number of annual deaths linked to cancer (around 30 000 deaths) according to the Institut National Du Cancer (INCA). It is a real public health issue, its incidence has been increasing above all in women and its prognosis is grim. The 1-year survival rate is 43% and 5-year survival rate 14% whatever the stage of the disease.

The Picardy region presents an excess mortality of 18% compared to the national average for the lung cancer and Somme has one of the highest incidence rate in France for this cancer.

Research hypothesis:

If the investigators know that tobacco smoke is the main risk factor, the other feature of this cancer is characterized by a diagnosis at an advanced stage when only limited, palliative treatments which are heavy, and costly can be provided Proposing the screening test with low dose helical computed tomography (LD-CT) has the aim to spot this cancer at an early stage when a curative surgical treatment is still possible in order to improve the survival chances.

Indeed screening by low dose CT showed a decrease of the death rate by 20 % of lung cancer and by 6 % for all the causes in the National Lung Screening Trial published in 2011.

If this screening test has for goal to diagnose lung cancers at an early stage, it also highlights in a quarter of the cases benign abnormalities requiring mainly further non invasive explorations. This low specificity is one of the reasons why in France the Haute Autorite Sante (HAS) has concluded that the current conditions were not met to authorize this screening in general population and insist on carrying the research for this screening.

Decreasing the number of false positives by selecting the targeted population and optimizing the decision algorithms would enable to improve the specificity of low dose CT as screening test of lung cancer.

Description of the intervention:

The rationale of this project is to use already existing networks among health care providers and between the health care providers and the departmental cancer screening agency (ADEMA 80) which is already in charge with the breast and colon cancer screening.

The targeted population of this screening concerns men and women from 55 to 74 year old who are smoking with a tobacco exposure of more than 30 pack-years or those who stopped for less than 15 years without obvious symptoms and who accept the screening tests with information on the results and the consequences which can arise ( non invasive exploration , CT after 3 months, Positon Emission Tomography scan or invasive exploration : CT guided biopsy, bronchoscopy, surgical exploration ) and who signed a consent form.

People with a history of cancer of less than 5 years, worsening of their health state, heart or respiratory morbidities which prevent a chest surgery are excluded of this study.

The population which is likely to undergo this test (male and female smokers from 55 to 74 years old) is estimated to 48 000 inhabitants for the department of the Somme which has a total population of 584 000 inhabitants.

The screening test is offered by primary care doctors and pneumologists of the Somme whom an invitation was sent by mail and who have accepted the way and means of the study.

The CT is prescribed on a prescription pad with 3 carbonless documents delivered by ADEMA 80 to the participating doctors: a part for the patient in order to take an appointment for his exam, one part which is sent back to ADEMA 80 with a prepaid envelope to keep a track and one part for the prescribing doctor. The LD-CT is carried out in radiology centers which comply with the charter of good practice of LD-CT.

The General Practitioners (GPs) and the pneumologists deal with the management of abnormalities which are eventually found by the CT according to the decision algorithms defined by the steering committee which has also validated a standard CT report. If the LD-CT proves to be normal, the screening is negative, the patient is invited again by ADEMA 80 the following year for a new LD-CT.

If the CT is abnormal , depending on the nodule' s size and/or nature either a new LD-CT is carried out after 3 months or if the screening is positive the patient's case is presented during a multidisciplinary team meeting with pneumologists, radiologists, oncologists, thoracic surgeons, pathologists.

Participants of the screening are being made aware of the benefits of quitting smoking and refer to a consultation on tobacco control if necessary.

A copy of the CT results is given to the local cancer screening agency (ADEMA 80) which is in charge with keeping a track and with statistic analyses.

This is a study with 2-year inclusion period. The length of the study is of 3 years.

It is the first study of lung cancer screening by LD-CT which is made at a regional scale in France.

Expected public health impact. The main objective of this screening is to assess the feasibility of an organized individual screening by LD-CT for a heavy smoker population aged from 55 to 74 in the Somme department, department with high incidence of lung cancer.

The secondary goals are to determine incidence of false positives, the number of screened cancers and staging, the histological subtypes, the sensibility and the specificity of this screening, to assess the treatments which have been implemented and the time it takes to deliver appropriate, to rate the quality of life and assess the incentive means to quit smoking

ELIGIBILITY:
Inclusion Criteria:

* male or female
* smokers or former smoker,
* aged between 55 and 74
* tobacco exposure of more than 30 pack-years,
* active smokers or who quitted for less than 15 years,
* obvious symptoms.

Exclusion Criteria:criteria:

* history of cancer within the last 5 years other than non melanoma skin cancer or carcinoma in situ,
* worsening of their health state with Eastern Cooperative Oncology Group performance status>3,-
* heart or respiratory severe co-morbidity with contraindications to thoracoscopy

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1307 (Estimated)
Dates: Start 2016-05-15 (Actual); Primary Completion 2020-05-15 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
feasibility of lung cancer screening implementation in France: participation rate | 3 years
  number of participants, participation rate : number of LD CT scan performed/ number of participants
efficacity of lung cancer screening in France: number of lung cancer diagnosed, number of stage I, rate of surgery, rate of false positive | 3 years
  number of lung cancer diagnosed, number of stage I, rate of surgery, rate of false positive

CONTACTS AND LOCATIONS:
Overall Officials: olivier LELEU, Principal Investigator — MD
Locations (1):
- LELEU, Abbeville, Somme, France

IPD SHARING:
Plan to Share IPD: Undecided